CLINICAL TRIAL: NCT04489407
Title: Can Remote Photoplethysmography Be Used for Contactless Vital Sign Acquisition in a Healthcare Setting? A Prospective Comparative Study.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lady Davis Institute (Other)
Collaborators: Carebook Technologies Inc. (Unknown)
Responsible Party: Principal Investigator, Noura Hassan, MD, MPH, FRCSC. Assistant Clinical Professor. Chair, Committee for Assessment of Medical Acts, Lady Davis Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-2376
Record Dates: First submitted 2020-07-23; First posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Coronavirus; Cardiac Disease; Respiratory Disease; Vascular Diseases
Keywords: oximetry; pulse oximetry; respiratory rate; remote photoplethysmography; coronavirus
MeSH Terms: conditions — Coronavirus Infections; Heart Diseases; Respiration Disorders; Vascular Diseases

STUDY DESIGN:
Intervention Model Description: Subjects enrolled in the study will be undergoing vital sign monitoring with the rPPG vital sign monitoring app and the conventional vital sign monitor. Readings with each vital sign monitoring technology will be taken simultaneously on all enrolled subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rPPG Vital Sign Monitor Readings (Experimental): Oxygen saturation, heart rate and respiratory rate obtained with the rPPG app.
  Interventions: Device: Remote Photoplethysmography (rPPG) vital sign acquisition
- Conventional Vital Sign Monitor Readings (Other): Oxygen saturation, heart rate and respiratory rate obtained with conventional vital sign monitors and manual respiratory rate counts.
  Interventions: Device: Remote Photoplethysmography (rPPG) vital sign acquisition

INTERVENTIONS:
Device: Remote Photoplethysmography (rPPG) vital sign acquisition — Subject vital signs will be acquired using the rPPG app simultaneously with the conventional vital sign monitors and manual respiratory rate calculation.
  Other Names: Welch Allyn Connex Vital Signs Monitor 6000 Series; Welch Allyn Vital Signs Monitor 7000 Series; Masimo Radical 7; Welch Allyn Vital Signs Monitor 6000 Series with Masimo rainbow SET Radical-7R pulse oximeter

SUMMARY:
Contactless and widely available health monitoring technologies are of growing interest in the context of the worldwide COVID-19 pandemic. Remote photoplethysmography (rPPG) is a well-studied technology that interprets variations in skin colour related to blood flow which, when analysed with complex mathematical algorithm, generates vital sign readings. This technology has been refined and embedded in a smartphone app designed to acquire heart rate, respiratory rate and oxygen saturation using a front-facing smartphone camera.

Preliminary data comparing the accuracy of smartphone rPPG readings with conventional vital sign monitor readings are promising; however, less than 5% of the population studied in the app development phase had oxygen saturation levels below 95% making it impossible to ensure reliability in these populations.

The goal of this study is to compare readings acquired using this rPPG app with the readings from hospital grade, Health Canada approved vital signs monitors used in healthcare settings with a focus on subject with low oxygen saturations. We will also study other sociodemographic and clinical features that may influence the accuracy of the readings. This will be achieved by recruiting consenting adults presenting to care in acute care settings and a designated COVID outpatient clinic. Vital signs will be acquired using the rPPG app and conventional hospital vital sign monitors simultaneously. Readings will be repeated within 2-5 minutes when time permits. Statistical analysis will be performed to analyze the findings and determine the accuracy and precision of the rPPG app readings.

It is expected that the vital sign readings acquired with the rPPG app will be almost identical to those acquired using hospital-grade monitors for all subjects regardless of age, gender, skin colour, COVID status and relevant comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Persons willing to participate and capable of providing informed consent, age of 18 years of more.
* Person able to sit still for the duration of the reading (maximum 2 minutes per reading).
* Persons with freckles, discreet skin pigmentation changes

Exclusion Criteria:

* Unable to provide informed consent
* Persons who are unable to follow basic instructions due to altered mental status, delirium, dementia or other conditions.
* Age < 18
* Intubated patients and patients requiring masks for supplemental oxygen
* Persons refusing to remove masks, eyewear, or clothing obstructing the face for the duration of readings.
* Persons with facial tattoos, large birthmarks or other skin alterations (scars, hemangiomas) on their nose or upper cheeks (cheekbones).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of rPPG heart rate | immediate; paired reading
  Accuracy of rPPG heart rate compared to conventional vital sign monitor heart rate readings. Comparison of each paired reading.
Accuracy of rPPG oxygen saturation | immediate; paired reading
  Accuracy of rPPG oxygen saturation compared to conventional vital sign monitor oxygen saturation readings. Comparison of discrepancy within each paired reading set.
Accuracy of rPPG respiratory rate | immediate; paired reading
  Accuracy of rPPG respiratory rate compared to manual counting of respiratory rate over 60 seconds. Comparison of discrepancy within each paired reading set.

SECONDARY OUTCOMES:
Reproducibility of rPPG heart rate readings | 2-5 minutes
  Comparison of rPPG heart rate results obtained on a given patient on serial readings within 2 minutes of each other.
Reproducibility of rPPG oxygen saturation readings | 2-5 minutes
  Comparison of rPPG oxygen saturation results obtained on a given patient on serial readings within 2 minutes of each other.
Reproducibility of rPPG respiratory rate readings | 2-5 minutes
  Comparison of rPPG respiratory rate results obtained on a given patient on serial readings within 2 minutes of each other.

OTHER OUTCOMES:
Accuracy of rPPG readings by oxygen saturation level | immediate; stratified analysis
  Analysis of accuracy of rPPG vital sign readings when stratified by oxygen saturation per conventional monitors stratified as follows: 95-100%; 90-94%; 85-89%; Less than 85%
Accuracy of rPPG readings by skin colour | immediate; stratified analysis
  Analysis of accuracy of rPPG vital sign readings when stratified by skin colour per the Fitzpatrick scale
Accuracy of rPPG readings by gender | immediate; stratified analysis
  Analysis of accuracy of rPPG vital sign readings when stratified for gender
Accuracy of rPPG readings by age | immediate; stratified analysis
  Analysis of accuracy of rPPG vital sign readings when stratified by age group
Accuracy of rPPG readings by comorbidity | immediate; stratified analysis
  Analysis of accuracy of rPPG vital sign readings when stratified for COVID, respiratory conditions, cardiac conditions and vascular conditions.

IPD SHARING:
Plan to Share IPD: No